CLINICAL TRIAL: NCT03725020
Title: Efficacy of a Novel Fluoride Varnish Formula in Preventing White Spot Lesions During and After Treatment With Fixed Orthodontic Appliances
Brief Title: Efficacy of a Novel Fluoride Varnish in Preventing WSL During/After Treatment With Fixed Orthodontic Appliances
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Malmö University (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Mikael Sonesson, Lecturer, Malmö University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MalmoUSonesson
Record Dates: First submitted 2018-10-29; First posted 2018-10-30 (Actual); Last update posted 2018-11-06 (Actual); Status verified 2018-11

CONDITIONS: Orthodontic Appliance Complication
Keywords: Orthodontics; Fixed appliance; White Spot Lesions; Fluoride varnish

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fluoride varnish (Experimental): During the course of the orthodontic treatment, the patients are regularly checked every 6th week. At the end of each such occasion, the clinical staff will apply the test varnish with a small brush in a thin layer around the base of the braces on the maxillary teeth. The varnish is let to dry and the subjects are instructed not to eat or drink within 60 minutes after the application. The NFV test varnish has mint flavour and the active ingredient is ammonium fluoride dissolved in ethanol, water and an acrylate polymer.
  Interventions: Other: Fluoride varnish
- Varnish without Fluoride (Placebo Comparator): During the course of the orthodontic treatment, the patients are regularly checked every 6th week. At the end of each such occasion, the clinical staff will apply either the placebo varnish with a small brush in a thin layer around the base of the braces on the maxillary teeth. The varnish is let to dry and the subjects are instructed not to eat or drink within 60 minutes after the application. The placebo varnish has an identical composition as the test varnish except for the ammonium fluoride. Thus, taste, colour and handling properties are the same.
  Interventions: Other: Fluoride varnish

INTERVENTIONS:
Other: Fluoride varnish — The study will employ a double-blind, randomized placebo-controlled design with two parallel groups. The intervention will start at onset of the fixed appliances and will be finalized one year after debond. The primary outcome will be incidence of white spot lesions on the labial surfaces of the maxillary incisors, canines and premolars, as assessed from high-resolution digital photos. The secondary outcome is the prevalence of WSLs at debonding.

SUMMARY:
The aim of the present study is to evaluate the efficacy of a novel fluoride varnish (NFV) in preventing white spot lesion development in adolescents during and after treatment with fixed orthodontic appliances.

DETAILED DESCRIPTION:
The study will employ a double-blind, randomized placebo-controlled design with two parallel groups. The intervention will start at onset of the fixed appliances and will be finalized one year after debonding. The primary outcome will be incidence of white spot lesions on the labial surfaces of the maxillary incisors, canines and premolars, as assessed from high-resolution digital photos. The secondary outcome is the prevalence of WSLs at debonding.

During the course of the orthodontic treatment, the patients are regularly checked every 6th week. At the end of each such occasion, the clinical staff will apply either the test or the placebo varnish with a small brush in a thin layer around the base of the braces on the maxillary teeth.

The pre- and post-treatment photos are projected on a screen (Hewlett Packard ProBook 6650b, Palo Alto CA, USA) in a dark room and the incidence and severity of enamel demineralization will be registered independently by two experienced and calibrated orthodontists according to the index of Gorelick et al. (1982).

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criterion is a scheduled treatment with fixed maxillary appliances according a standard straight-wire concept (McLaughlin et al., 2001) during a period of at least 12 months

Exclusion Criteria:

* In the event of long-term prescriptions of general antibiotics during the course of the study, this should be recorded separately

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 180 (Actual)
Dates: Start 2014-06-01 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
The primary outcome will be incidence of white spot lesions on the labial surfaces of the maxillary incisors, canines and premolars | 12-24 months
  Assessed from high-resolution digital photos

SECONDARY OUTCOMES:
The secondary outcome is the prevalence of WSLs at debonding and one year after debond | 12 months
  Assessed from high-resolution digital photos

CONTACTS AND LOCATIONS:
Overall Officials: Mikael Sonesson, Odont. Dr., Principal Investigator — Malmö University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sonesson M, Brechter A, Lindman R, Abdulraheem S, Twetman S. Fluoride varnish for white spot lesion prevention during orthodontic treatment: results of a randomized controlled trial 1 year after debonding. Eur J Orthod. 2021 Aug 3;43(4):473-477. doi: 10.1093/ejo/cjaa055. PMID 33009565
- [Derived] Sonesson M, Brechter A, Abdulraheem S, Lindman R, Twetman S. Fluoride varnish for the prevention of white spot lesions during orthodontic treatment with fixed appliances: a randomized controlled trial. Eur J Orthod. 2020 Jun 23;42(3):326-330. doi: 10.1093/ejo/cjz045. PMID 31197364